CLINICAL TRIAL: NCT00740636
Title: Phase II Study of Temozolomide for Relapsed Sensitive or Refractory Small Cell Lung Cancer
Brief Title: Temozolomide for Relapsed Sensitive or Refractory Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-065
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-06

CONDITIONS: Lung Cancer
Keywords: TEMOZOLOMIDE; Lung
MeSH Terms: conditions — Lung Neoplasms | interventions — Temozolomide

ARMS (2):
- 75 mg/m2/day Temozolomide (Experimental): 75 mg/m2/day Temozolomide for 21 days (7 days off treatment). 28 day cycles.
  Interventions: Drug: Temozolomide
- 200 mg/m2/day Temozolomide (Experimental): 200 mg/m2/day Temozolomide for 5 days (23 days off treatment). 28 day cycles.
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Temozolomide — Temozolomide will be administered orally once per day on days 1 through 5 of a 28 day cycle. The dose will be 75 mg/m2/day.
  Arms: 75 mg/m2/day Temozolomide
Drug: Temozolomide — Temozolomide will be administered orally once per day on days 1 through 5 of a 28 day cycle. The dose will be 200mg/m2/day.
  Arms: 200 mg/m2/day Temozolomide

SUMMARY:
The purpose of this study is to determine whether treatment with temozolomide will shrink small cell lung cancer tumors. Temozolomide is an oral chemotherapy drug that is currently used to treat brain cancer and melanoma.

As part of this study, we will be doing additional tests that may help us understand how temozolomide works. First, if there is a tumor sample from a biopsy done in the past, it will be analyzed for an abnormal gene that may be present in lung cancer. Before starting temozolomide, a research blood test will be done to look for the same abnormal gene we are looking for in your tumor sample. Also, before starting temozolomide and every time you have a repeat CT scan, a research blood test will be done to analyze the number of tumor cells in your bloodstream.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed SCLC at MSKCC that has progressed after one or two chemotherapy regimens.
* At least 3 weeks must have elapsed since last chemotherapy or radiation treatment and initiation of study treatment.
* Karnofsky performance status > or = to 60%.
* Patients must have measurable disease, this can include brain metastases.
* Patients must have normal organ and marrow function as defined below:
* - leukocytes > 3,000/mcL
* platelets > 100,000/mcL
* total bilirubin < 1.5 mg/dL
* AST(SGOT)/ALT(SGPT) < 2.5 X institutional upper limit of normal
* Creatinine < 2.0 mg/dl
* For women of child-bearing potential, negative pregnancy test within 7 days prior to starting temozolomide.
* Men and women of childbearing potential must agree to practice adequate contraception.
* Ability to understand and the willingness to sign a written informed consent document.
* Both men and women of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

* Patients who have not recovered from adverse events of previous therapies.
* Patients receiving other investigational agents.
* Patients with leptomeningeal involvement.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements.
* Acquired Immune Deficiency Syndrome (AIDS) based upon current CDC definition or HIV-positive patients on combination antiretroviral therapy. However, HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because these patients are at increased risk of lethal infections when treated with marrow- suppressive therapy. Excluding patients on HAART is necessary due to the potential for pharmacokinetic interactions with temozolomide.
* Women who are pregnant or breast feeding, due to possible adverse effects on the developing fetus or infant due to study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Pietanza, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - Memoral Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center@Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- 200 mg/m2/Day for 5 Days (23 Days Off tx). 28 Day Cycles.: 200 mg/m2/day for 5 days (23 days off treatment). 28 day cycles.
- 75 mg/m2/Day for 21 Days (7 Days Off tx). 28 Day Cycles.: 75 mg/m2/day for 21 days (7 days off treatment). 28 day cycles.
Period: Overall Study
Arm/Group | 200 mg/m2/Day for 5 Days (23 Days Off tx). 28 Day Cycles. | 75 mg/m2/Day for 21 Days (7 Days Off tx). 28 Day Cycles.
Started | 25 | 67
Completed | 23 | 63
Not Completed | 2 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Patient Ineligible | 0 | 1
Not completed — Patient Not Treated | 0 | 1
Not completed — Progressive Disease | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 200 mg/m2/Day for 5 Days (23 Days Off tx). 28 Day Cycles. | 75 mg/m2/Day for 21 Days (7 Days Off tx). 28 Day Cycles. | Total
Number analyzed (Participants) | 25 | 67 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 22 | 36
  >=65 years | 11 | 45 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 37 | 53
  Male | 9 | 30 | 39

OUTCOME MEASURES:

1. Primary Outcome: The Objective Overall Response
Description: The objective response is defined as all complete responses and partial responses based on the modified RECIST.Complete Response (CR): Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | 200 mg/m2/Day for 5 Days (23 Days Off tx). 28 Day Cycles. | 75 mg/m2/Day for 21 Days (7 Days Off tx). 28 Day Cycles.
Number analyzed (Participants) | 23 | 63
participants
  Partial Response (PR) | 7 | 12
  Stable Disease (SD) | 7 | 19
  Progression of Disease (POD) | 9 | 31
  Complete Response (CR) | 0 | 1

ADVERSE EVENTS:
Arm/Group | 200 mg/m2/Day for 5 Days (23 Days Off tx). 28 Day Cycles. | 75 mg/m2/Day for 21 Days (7 Days Off tx). 28 Day Cycles.
Serious Adverse Events (participants affected / at risk) | 12/25 | 20/67
Other Adverse Events (participants affected / at risk) | 20/25 | 51/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg/m2/Day for 5 Days (23 Days Off tx). 28 Day Cycles. (N=25) | 75 mg/m2/Day for 21 Days (7 Days Off tx). 28 Day Cycles. (N=67)
Death not assoc w CTCAE term- Death NOS (General disorders) | 1 (1) | 0 (0)
Death not assoc w CTCAE term-Disease prog NOS (General disorders) | 3 (3) | 1 (1)
Dehydration (General disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 1 (1) | 3 (3)
Infection w/ Gr 3/4 neut, Lung (pneumonia) (Infections and infestations) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (4) | 3 (3)
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Somnolence/depressed level of conscious (General disorders) | 1 (1) | 0 (0)
Thrombosis/thrombus/embolism (Cardiac disorders) | 2 (2) | 0 (0)
AST, SGOT (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ataxia (incoordination) (Nervous system disorders) | 0 (0) | 1 (1)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 2 (2)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Edema: limb (General disorders) | 0 (0) | 2 (2)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hemorrhage/Bleeding, other (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypoxia (General disorders) | 0 (0) | 2 (2)
Inf norm ANC/gr1/2 neut-Pneumonia(lung) (Infections and infestations) | 0 (0) | 2 (2)
Infection unknown ANC-UTI NOS (Infections and infestations) | 0 (0) | 1 (1)
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Neurology - Other (Nervous system disorders) | 0 (0) | 1 (1)
Potassium, low (hypokalemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Secondary malignancy possibly related to treatment (General disorders) | 0 (0) | 1 (1)
Secondary malig-poss related to ca txt specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 1 (1)
Muscle weakness - Whole body/general (General disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 200 mg/m2/Day for 5 Days (23 Days Off tx). 28 Day Cycles. (N=25) | 75 mg/m2/Day for 21 Days (7 Days Off tx). 28 Day Cycles. (N=67)
Constipation (Gastrointestinal disorders) | 5 (5) | 7 (7)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (11)
ALT, SGPT (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
AST, SGOT (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (7)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 6 (8) | 21 (34)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 2 (2) | 14 (14)
Hemoglobin (Blood and lymphatic system disorders) | 5 (5) | 17 (17)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 6 (6) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 6 (6) | 26 (26)
Nausea (General disorders) | 2 (4) | 9 (9)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Pain - Head/headache (General disorders) | 2 (2) | 0 (0)
Pain - Other (General disorders) | 2 (3) | 0 (0)
Phosphate, low (hypophosphatemia) (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 6 (6) | 5 (5)
Sodium, low (hyponatremia) (Metabolism and nutrition disorders) | 2 (2) | 8 (8)
Vomiting (General disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes